CLINICAL TRIAL: NCT05194124
Title: A Phase 3, Randomized, Double-Blind Trial of Two Formulations of Setmelanotide (Daily and Weekly) With a Crossover to Open-Label Once Weekly Setmelanotide in Patients With Specific Gene Defects in the Melanocortin-4 Receptor Pathway Who Are Currently on a Stable Dose of the Once Daily Formulation
Brief Title: Phase 3 Crossover Trial of Two Formulations of Setmelanotide in Participants With Specific Gene Defects in the MC4R Pathway
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-037
Record Dates: First submitted 2021-07-27; First posted 2022-01-18 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Bardet-Biedl Syndrome; POMC Deficiency
Keywords: Melanocortin-4 Receptor Pathway; Genetic Obesity; Hunger; Hyperphagia
MeSH Terms: conditions — Bardet-Biedl Syndrome; Proopiomelanocortin Deficiency; Hyperphagia | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Run-in Period: Setmelanotide 2 mg QD (Experimental): Participants received subcutaneous (SC) injection of 2 mg setmelanotide once daily (QD) for 1 week in the run-in period.
  Interventions: Drug: Setmelanotide 2 mg
- Run-in Period: Setmelanotide 2.5 mg QD (Experimental): Participants received SC injection of 2.5 mg setmelanotide QD for 1 week in the run-in period.
  Interventions: Drug: Setmelanotide 2.5 mg
- Run-in Period: Setmelanotide 3 mg QD (Experimental): Participants received SC injection of 3 mg setmelanotide QD for 1 week in the run-in period.
  Interventions: Drug: Setmelanotide 3 mg
- DB Period: Setmelanotide 20 mg QW (Experimental): Participants who received 2 mg setmelanotide QD in the run-in period, received SC injection of 20 mg setmelanotide once weekly (QW) and placebo matched to setmelanotide QD for 13 weeks in the DB period.
  Interventions: Drug: Setmelanotide 20 mg
- DB Period: Setmelanotide 25 mg QW (Experimental): Participants who received 2.5 mg setmelanotide QD in the run-in period, received SC injection of 25 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks in the DB period.
  Interventions: Drug: Setmelanotide 25 mg
- DB Period: Setmelanotide 3 mg QD (Experimental): Participants who received 3 mg setmelanotide QD in the run-in period, received SC injection of 3 mg setmelanotide QD and placebo matched to setmelanotide QW for 13 weeks in the DB period.
  Interventions: Drug: Setmelanotide 3 mg
- DB Period: Setmelanotide 30 mg QW (Experimental): Participants who received 3 mg setmelanotide QD in the run-in period, received SC injection of 30 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks in the DB period.
  Interventions: Drug: Setmelanotide 30 mg
- OL Period: Setmelanotide 20 mg QW (Experimental): Participants who received 2 mg setmelanotide QD in the run-in period and 20 mg setmelanotide QW in the DB period, received SC injection of 20 mg setmelanotide QW for 13 weeks in the OL period.
  Interventions: Drug: Setmelanotide 20 mg
- OL Period: Setmelanotide 25 mg QW (Experimental): Participants who received 2.5 mg setmelanotide QD in the run-in period and 25 mg setmelanotide QW in the DB period, received SC injection of 25 mg setmelanotide QW for 13 weeks in the OL period.
  Interventions: Drug: Setmelanotide 25 mg
- OL Period: Setmelanotide 30 mg QW (Experimental): Participants who received 3 setmelanotide QD in the run-in period and 3 mg setmelanotide QD or 30 mg setmelanotide QW in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
  Interventions: Drug: Setmelanotide 30 mg

INTERVENTIONS:
Drug: Setmelanotide 2 mg — Administered as SC injection
  Arms: Run-in Period: Setmelanotide 2 mg QD
Drug: Setmelanotide 2.5 mg — Administered as SC injection
  Arms: Run-in Period: Setmelanotide 2.5 mg QD
Drug: Setmelanotide 3 mg — Administered as SC injection
  Arms: DB Period: Setmelanotide 3 mg QD; Run-in Period: Setmelanotide 3 mg QD
Drug: Setmelanotide 20 mg — Administered as SC injection
  Arms: DB Period: Setmelanotide 20 mg QW; OL Period: Setmelanotide 20 mg QW
Drug: Setmelanotide 25 mg — Administered as SC injection
  Arms: DB Period: Setmelanotide 25 mg QW; OL Period: Setmelanotide 25 mg QW
Drug: Setmelanotide 30 mg — Administered as SC injection
  Arms: DB Period: Setmelanotide 30 mg QW; OL Period: Setmelanotide 30 mg QW

SUMMARY:
A trial to compare the weekly and daily formulations of setmelanotide in participants with genetic defects in the melanocortin-4 receptor pathway.

DETAILED DESCRIPTION:
This study is designed to compare the safety, pharmacokinetics, and efficacy of weekly and daily formulations of setmelanotide in participants with obesity associated with biallelic or heterozygous POMC (pro-opiomelanocortin), PCSK1 (proprotein convertase subtilisin/kexin Type 1), LEPR (leptin receptor) genetic variants, and participants with Bardet-Biedl Syndrome (BBS).

ELIGIBILITY:
Key Inclusion Criteria:

* Biallelic or heterozygous POMC/PCSK1 or LEPR (PPL) genetic variants or Bardet-Biedl syndrome (BBS), for which they are being treated with QD setmelanotide.
* 6 years or older at screening.
* Taking the setmelanotide QD formulation for at least 6 months in the RM-493-022 (NCT03013543) study with acceptable safety and tolerability, and dose level.
* Participant and/or parent or guardian is able to communicate well with the Investigator, to understand and comply with the requirements of the study and is able to understand and sign the written informed consent/assent.
* Use of a highly effective form of contraception throughout the study and for 90 days following the study.

Key Exclusion Criteria:

* Glycosylated hemoglobin (HbA1C) >9.0% at screening.
* Anti-obesity medications within 3 months prior to starting the Run-in Period.
* History of significant liver disease or liver injury.
* Glomerular filtration rate <30 milliliter per minute (mL/min).
* Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions.
* Major psychiatric disorders.
* Any suicidal ideation or behavior, or any lifetime history of a suicide attempt.
* Significant hypersensitivity to any excipient in the study drug.
* Inability to comply with the QW and QD injection regimens.
* Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing, with the exception of a setmelanotide clinical trial.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (7):
- United States (2):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin
- Alberta Health Services, Edmonton, Alberta, Canada
- Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin, Germany
- Erasmus MC, Rotterdam, Netherlands
- UPR Medical Sciences Campus, Rio Piedras, Puerto Rico
- Addenbrooke's Hospital, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were screened and 19 were randomized and treated in this study. The study consisted of a run-in period of up to 1 week in which the participants received once daily (QD) setmelanotide [2 milligrams (mg), 2.5 mg, or 3 mg]; a 13-week double-blind period in which the participants were randomized to either QD or once weekly (QW) setmelanotide; and a 13-week non-randomized open-label period where all participants received open label QW setmelanotide.
Groups:
- Run-in Period: Setmelanotide 2 mg QD: Participants received subcutaneous (SC) injection of 2 mg setmelanotide QD for 1 week in the run-in period.
- DB Period: Setmelanotide 20 mg QW: Participants who received 2 mg setmelanotide QD in the run-in period, received SC injection of 20 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks in the DB period.
Period: Run-in Period (1 Week)
Arm/Group | Run-in Period: Setmelanotide 2 mg QD | Run-in Period: Setmelanotide 2.5 mg QD | Run-in Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 20 mg QW | DB Period: Setmelanotide 25 mg QW | DB Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 30 mg QW | OL Period: Setmelanotide 20 mg QW | OL Period: Setmelanotide 25 mg QW | OL Period: Setmelanotide 30 mg QW
Started | 2 | 1 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double Blind (DB) Period (13 Weeks)
Arm/Group | Run-in Period: Setmelanotide 2 mg QD | Run-in Period: Setmelanotide 2.5 mg QD | Run-in Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 20 mg QW | DB Period: Setmelanotide 25 mg QW | DB Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 30 mg QW | OL Period: Setmelanotide 20 mg QW | OL Period: Setmelanotide 25 mg QW | OL Period: Setmelanotide 30 mg QW
Started | 0 | 0 | 0 | 2 | 1 | 9 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 1 | 7 | 7 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Period: Open Label (OL) Period (13 Weeks)
Arm/Group | Run-in Period: Setmelanotide 2 mg QD | Run-in Period: Setmelanotide 2.5 mg QD | Run-in Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 20 mg QW | DB Period: Setmelanotide 25 mg QW | DB Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 30 mg QW | OL Period: Setmelanotide 20 mg QW | OL Period: Setmelanotide 25 mg QW | OL Period: Setmelanotide 30 mg QW
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 14 (7 participants from DB Phase: Setmelanotide 3 mg QD group and 7 participants from DB Phase: Setmelanotide 3 mg QW group)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of setmelanotide after the randomization.
Groups:
- Setmelanotide 2 mg QD: Run-in Period: Participants received SC injection of 2 mg setmelanotide QD for 1 week.
  DB Period: Participants received SC injection of 20 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks.
  OL Period: Participants received SC injection of 20 mg setmelanotide QW for 13 weeks.
- Setmelanotide 2.5 mg QD: Run-in Period: Participants received SC injection of 2.5 mg setmelanotide QD for 1 week.
  DB Period: Participants received SC injection of 25 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks.
  OL Period: Participants received SC injection of 25 mg setmelanotide QW for 13 weeks.
- Setmelanotide 3 mg QD: Run-in Period: Participants received SC injection of 3 mg setmelanotide QD for 1 week.
  DB Period: Participants received SC injection of 3 mg setmelanotide QD and placebo matched to setmelanotide QW or 30 mg setmelanotide QW and placebo matched to setmelanotide QD for 13 weeks.
  OL Period: Participants received SC injection of 30 mg setmelanotide QW for 13 weeks.
- Total: Total of all reporting groups
Arm/Group | Setmelanotide 2 mg QD | Setmelanotide 2.5 mg QD | Setmelanotide 3 mg QD | Total
Number analyzed (Participants) | 2 | 1 | 16 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (12.73) | 19.0 | 20.8 (8.30) | 20.6 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 10 | 11
  Male | 2 | 0 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 2 | 1 | 14 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 0 | 1
  Race: White | 1 | 1 | 14 | 16
  Race: Other | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration (Cmax) of Setmelanotide After QD Administration in the Run-in Period
Description: Maximum drug concentration determined directly from individual concentration-time data.
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose at Week -1
Population: Participants in the Pharmacokinetic Analysis Set (PKAS) (all participants who received at least 1 dose of setmelanotide and who had a sufficient number of measurable plasma concentrations to permit assessment of noncompartmental parameters) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Setmelanotide 2 mg QD: Participants received SC injection of 2 mg setmelanotide QD for 1 week.
- Setmelanotide 2.5 mg QD: Participants received SC injection of 2.5 mg setmelanotide QD for 1 week.
- Setmelanotide 3 mg QD: Participants received SC injection of 3 mg setmelanotide QD for 1 week.
Arm/Group | Setmelanotide 2 mg QD | Setmelanotide 2.5 mg QD | Setmelanotide 3 mg QD
Number analyzed (Participants) | 2 | 1 | 16
nanograms per milliliter (ng/mL) | 29.4 (3.49) | 44.8 | 59.9 (29.6)

2. Primary Outcome: Cmax of Setmelanotide After QW Administration
Description: Maximum drug concentration determined directly from individual concentration-time data. Data are reported by dose level (treatment regimen) in the OL Period and dosing sequence (QD-QD-QW or QD-QW-QW).
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours postdose at Week 14
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Setmelanotide 20 mg QW (QD-QW-QW): Participants who received 2 mg setmelanotide QD in the run-in period and 20 mg setmelanotide QW in the DB period, received SC injection of 20 mg setmelanotide QW for 13 weeks in the OL period.
- Setmelanotide 25 mg QW (QD-QW-QW): Participants who received 2.5 mg setmelanotide QD in the run-in period and 25 mg setmelanotide QW in the DB period, received SC injection of 25 mg setmelanotide QW for 13 weeks in the OL period.
- Setmelanotide 30 mg QW (QD-QD-QW): Participants who received 3 mg setmelanotide QD in the run-in period and 3 mg setmelanotide QD in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
- Setmelanotide 30 mg QW (QD-QW-QW): Participants who received 3 mg setmelanotide QD in the run-in period and 30 mg setmelanotide QW in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 30 mg QW (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 7 | 7
ng/mL | 22.4 | 32.7 | 31.8 (28.6) | 57.3 (33.0)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Setmelanotide After QD Administration in the Run-in Period
Description: Maximum drug concentration determined directly from individual concentration-time data.
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose at Week -1
Population: Participants in the PKAS with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Setmelanotide 2 mg QD | Setmelanotide 2.5 mg QD | Setmelanotide 3 mg QD
Number analyzed (Participants) | 2 | 1 | 16
hours | 6.91 [5.92 to 7.90] | 5.88 | 6.02 [2.00 to 8.00]

4. Primary Outcome: Tmax of Setmelanotide After QW Administration
Description: as for outcome 2
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours postdose at Week 14
Population: Participants in the PKAS with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 30 mg QW (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 7 | 7
hours | 3.93 | 5.93 | 1.98 [0.500 to 6.00] | 5.95 [2.03 to 6.03]

5. Primary Outcome: Mean Trough Plasma Concentration (Ctrough) of Setmelanotide After QD or QW Administration at Week 1
Description: Ctrough is concentration at the end of the dosing interval, prior to subsequent dose administration. Data are reported by dose level (treatment regimen) in the DB Period and dosing sequence (QD-QD-QW or QD-QW-QW).
Time Frame: 30 minutes predose at Week 1
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Setmelanotide 3 mg QD (QD-QD-QW): Participants who received 3 mg setmelanotide QD in the run-in period and 3 mg setmelanotide QD in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 2 | 1 | 9 | 7
ng/mL | 5.17 (0.856) | 4.36 | 11.7 (13.5) | 16.6 (16.3)

6. Primary Outcome: Mean Setmelanotide Ctrough After QD or QW Administration at Week 5
Description: as for outcome 5
Time Frame: 30 minutes predose at Week 5
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 0 | 1 | 7 | 7
ng/mL |  | 9.54 | 12.2 (7.62) | 15.6 (13.3)

7. Primary Outcome: Mean Setmelanotide Ctrough After QD or QW Administration at Week 9
Description: as for outcome 5
Time Frame: 30 minutes predose at Week 9
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 7 | 6
ng/mL | 11.1 | 6.43 | 12.3 (11.4) | 20.1 (13.7)

8. Primary Outcome: Mean Setmelanotide Ctrough After QD or QW Administration at Week 18
Description: as for outcome 5
Time Frame: 30 minutes predose at Week 18
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 6 | 6
ng/mL | 14.4 | 12.6 | 13.6 (13.9) | 26.2 (23.8)

9. Primary Outcome: Mean Setmelanotide Ctrough After QD or QW Administration at Week 22
Description: as for outcome 5
Time Frame: 30 minutes predose at Week 22
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 6 | 7
ng/mL | 11.9 | 14.3 | 17.0 (15.4) | 27.9 (25.4)

10. Primary Outcome: Mean Setmelanotide Ctrough After QD or QW Administration at Week 27
Description: as for outcome 5
Time Frame: 30 minutes predose at Week 27
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 3 mg QD (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 6 | 7
ng/mL | 14.2 | 9.91 | 20.3 (19.4) | 32.1 (23.9)

11. Primary Outcome: Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUC0-tau) of Setmelanotide After QD Administration in the Run-in Period
Description: AUC0-tau was recorded from collected blood samples.
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 6, and 8 hours postdose at Week -1
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Setmelanotide 2 mg QD | Setmelanotide 2.5 mg QD | Setmelanotide 3 mg QD
Number analyzed (Participants) | 0 | 0 | 7
hours*ng/mL |  |  | 975 (659)

12. Primary Outcome: AUC0-tau of Setmelanotide After QD Administration in the Run-in Period
Description: AUC0-tau was recorded from collected blood samples. Data are reported by dose level (treatment regimen) in the OL Period and dosing sequence (QD-QD-QW or QD-QW-QW).
Time Frame: Pre-dose (0 hour) and 0.5, 1, 2, 6, 8, 12, 24, 48, 72, 96, 120, and 168-hours postdose at Week 14
Population: Participants in the PKAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours*mg/mL
Arm/Group | Setmelanotide 20 mg QW (QD-QW-QW) | Setmelanotide 25 mg QW (QD-QW-QW) | Setmelanotide 30 mg QW (QD-QD-QW) | Setmelanotide 30 mg QW (QD-QW-QW)
Number analyzed (Participants) | 1 | 1 | 6 | 6
hours*mg/mL | 1590 | 2260 | 2470 (2890) | 5010 (4000)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The AEs reported after the start of the run-in period were considered TEAEs.
Time Frame: From first dose of study drug administration up to Week 30
Population: Participants in the Safety Analysis Set (all participants who received at least 1 dose of protocol-specified study drug) were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Period: Setmelanotide 2 mg QD: Participants received SC injection of 2 mg setmelanotide QD for 1 week in the run-in period.
Arm/Group | Run-in Period: Setmelanotide 2 mg QD | Run-in Period: Setmelanotide 2.5 mg QD | Run-in Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 20 mg QW | DB Period: Setmelanotide 25 mg QW | DB Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 30 mg QW | OL Period: Setmelanotide 20 mg QW | OL Period: Setmelanotide 25 mg QW | OL Period: Setmelanotide 30 mg QW
Number analyzed (Participants) | 2 | 1 | 16 | 2 | 1 | 9 | 7 | 1 | 1 | 14
Participants | 0 | 0 | 1 | 2 | 1 | 9 | 6 | 0 | 1 | 10

14. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) From Baseline Through Week 13
Description: The injection site evaluation included the identification of areas of erythema, edema, and induration, as well as the presence of localized pain, tenderness, and itching. Baseline was defined as the last available measurement prior to the first dose of setmelanotide or placebo. Injection site reactions frequency of once daily (QD) and once weekly (QW) were reported. Data are reported by dose level (treatment regimen) in the DB Period. Number of participants with injection site reactions according to severity were reported.
Time Frame: Baseline through Week 13
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Setmelanotide 20 mg QW: Participants who received 2 mg setmelanotide QD in the run-in period, received 20 mg setmelanotide QW in the DB period.
- Setmelanotide 25 mg QW: Participants who received 2.5 mg setmelanotide QD in the run-in period, received 25 mg setmelanotide QW in the DB period.
- Setmelanotide 3 mg QD: Participants who received 3 mg setmelanotide QD in the run-in period, received 3 mg setmelanotide QD in the DB period.
- Setmelanotide 30 mg QW: Participants who received 3 mg setmelanotide QD in the run-in period, received 30 mg setmelanotide QW in the DB period.
Arm/Group | Setmelanotide 20 mg QW | Setmelanotide 25 mg QW | Setmelanotide 3 mg QD | Setmelanotide 30 mg QW
Number analyzed (Participants) | 2 | 1 | 9 | 7
Participants
  Erythema QD: None | 2 | 0 | 7 | 5
  Erythema QD: Mild | 0 | 1 | 2 | 2
  Erythema QD: Moderate | 0 | 0 | 0 | 0
  Erythema QD: Severe | 0 | 0 | 0 | 0
  Erythema QW: None | 1 | 0 | 4 | 3
  Erythema QW: Mild | 1 | 1 | 4 | 3
  Erythema QW: Moderate | 0 | 0 | 1 | 1
  Erythema QW: Severe | 0 | 0 | 0 | 0
  Edema QD: None | 2 | 1 | 9 | 7
  Edema QD: Mild | 0 | 0 | 0 | 0
  Edema QD: Moderate | 0 | 0 | 0 | 0
  Edema QD: Severe | 0 | 0 | 0 | 0
  Edema QW: None | 2 | 1 | 9 | 6
  Edema QW: Mild | 0 | 0 | 0 | 1
  Edema QW: Moderate | 0 | 0 | 0 | 0
  Edema QW: Severe | 0 | 0 | 0 | 0
  Induration QD: None | 1 | 1 | 9 | 6
  Induration QD: Mild | 1 | 0 | 0 | 0
  Induration QD: Moderate | 0 | 0 | 0 | 1
  Induration QD: Severe | 0 | 0 | 0 | 0
  Induration QW: None | 1 | 0 | 8 | 4
  Induration QW: Mild | 1 | 1 | 1 | 2
  Induration QW: Moderate | 0 | 0 | 0 | 1
  Induration QW: Severe | 0 | 0 | 0 | 0
  Itching QD: None | 2 | 1 | 8 | 3
  Itching QD: Mild | 0 | 0 | 1 | 4
  Itching QD: Moderate | 0 | 0 | 0 | 0
  Itching QD: Severe | 0 | 0 | 0 | 0
  Itching QW: None | 2 | 1 | 9 | 2
  Itching QW: Mild | 0 | 0 | 0 | 4
  Itching QW: Moderate | 0 | 0 | 0 | 1
  Itching QW: Severe | 0 | 0 | 0 | 0
  Pain or Tenderness QD: None | 2 | 0 | 6 | 5
  Pain or Tenderness QD: Mild | 0 | 1 | 3 | 2
  Pain or Tenderness QD: Moderate | 0 | 0 | 0 | 0
  Pain or Tenderness QD: Severe | 0 | 0 | 0 | 0
  Pain or Tenderness QW: None | 2 | 0 | 6 | 1
  Pain or Tenderness QW: Mild | 0 | 1 | 3 | 2
  Pain or Tenderness QW: Moderate | 0 | 0 | 0 | 4
  Pain or Tenderness QW: Severe | 0 | 0 | 0 | 0
  Other QD: None | 1 | 1 | 9 | 7
  Other QD: Mild | 1 | 0 | 0 | 0
  Other QD: Moderate | 0 | 0 | 0 | 0
  Other QD: Severe | 0 | 0 | 0 | 0
  Other QW: None | 0 | 1 | 6 | 5
  Other QW: Mild | 2 | 0 | 3 | 1
  Other QW: Moderate | 0 | 0 | 0 | 1
  Other QW: Severe | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With ISRs From Week 14 Through Week 27
Description: The injection site evaluation included the identification of areas of erythema, edema, and induration, as well as the presence of localized pain, tenderness, and itching. Injection site reactions frequency of QD and QW were reported. Data are reported by dose level (treatment regimen) in the OL Period. Number of participants with injection site reactions according to severity were reported.
Time Frame: Week 14 through Week 27
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Setmelanotide 20 mg QW: Participants who received 2 mg setmelanotide QD in the run-in period and 20 mg setmelanotide QW in the DB period, received SC injection of 20 mg setmelanotide QW for 13 weeks in the OL period.
- Setmelanotide 25 mg QW: Participants who received 2.5 mg setmelanotide QD in the run-in period and 25 mg setmelanotide QW in the DB period, received SC injection of 25 mg setmelanotide QW for 13 weeks in the OL period.
- Setmelanotide 30 mg QW: Participants who received 3 mg setmelanotide QD in the run-in period and 3 mg setmelanotide QD or 30 mg setmelanotide QW in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
Arm/Group | Setmelanotide 20 mg QW | Setmelanotide 25 mg QW | Setmelanotide 30 mg QW
Number analyzed (Participants) | 1 | 1 | 14
Participants
  Erythema QD: None | 1 | 1 | 13
  Erythema QD: Mild | 0 | 0 | 1
  Erythema QD: Moderate | 0 | 0 | 0
  Erythema QD: Severe | 0 | 0 | 0
  Erythema QW: None | 1 | 0 | 12
  Erythema QW: Mild | 0 | 1 | 2
  Erythema QW: Moderate | 0 | 0 | 0
  Erythema QW: Severe | 0 | 0 | 0
  Edema QD: None | 1 | 1 | 13
  Edema QD: Mild | 0 | 0 | 1
  Edema QD: Moderate | 0 | 0 | 0
  Edema QD: Severe | 0 | 0 | 0
  Edema QW: None | 1 | 1 | 14
  Edema QW: Mild | 0 | 0 | 0
  Edema QW: Moderate | 0 | 0 | 0
  Edema QW: Severe | 0 | 0 | 0
  Induration QD: None | 1 | 1 | 13
  Induration QD: Mild | 0 | 0 | 1
  Induration QD: Moderate | 0 | 0 | 0
  Induration QD: Severe | 0 | 0 | 0
  Induration QW: None | 0 | 0 | 8
  Induration QW: Mild | 1 | 1 | 4
  Induration QW: Moderate | 0 | 0 | 2
  Induration QW: Severe | 0 | 0 | 0
  Itching QD: None | 1 | 1 | 14
  Itching QD: Mild | 0 | 0 | 0
  Itching QD: Moderate | 0 | 0 | 0
  Itching QD: Severe | 0 | 0 | 0
  Itching QW: None | 1 | 1 | 10
  Itching QW: Mild | 0 | 0 | 4
  Itching QW: Moderate | 0 | 0 | 0
  Itching QW: Severe | 0 | 0 | 0
  Pain or Tenderness QD: None | 1 | 1 | 13
  Pain or Tenderness QD: Mild | 0 | 0 | 1
  Pain or Tenderness QD: Moderate | 0 | 0 | 0
  Pain or Tenderness QD: Severe | 0 | 0 | 0
  Pain or Tenderness QW: None | 1 | 1 | 8
  Pain or Tenderness QW: Mild | 0 | 0 | 6
  Pain or Tenderness QW: Moderate | 0 | 0 | 0
  Pain or Tenderness QW: Severe | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to week 30
Description: Safety Analysis Set included all participants who received at least 1 dose of protocol-specified study drug.
Groups:
- OL Period: Setmelanotide 30 mg QW: Participants who received 3 setmelanotide QD in the run-in period and 30 mg setmelanotide QD or QW in the DB period, received SC injection of 30 mg setmelanotide QW for 13 weeks in the OL period.
Arm/Group | Run-in Period: Setmelanotide 2 mg QD | Run-in Period: Setmelanotide 2.5 mg QD | Run-in Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 20 mg QW | DB Period: Setmelanotide 25 mg QW | DB Period: Setmelanotide 3 mg QD | DB Period: Setmelanotide 30 mg QW | OL Period: Setmelanotide 20 mg QW | OL Period: Setmelanotide 25 mg QW | OL Period: Setmelanotide 30 mg QW
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/16 | 0/2 | 0/1 | 0/9 | 0/7 | 0/1 | 0/1 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/16 | 0/2 | 0/1 | 0/9 | 0/7 | 0/1 | 0/1 | 0/14
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 1/16 | 2/2 | 1/1 | 9/9 | 6/7 | 0/1 | 1/1 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Setmelanotide 2 mg QD (N=2) | Run-in Period: Setmelanotide 2.5 mg QD (N=1) | Run-in Period: Setmelanotide 3 mg QD (N=16) | DB Period: Setmelanotide 20 mg QW (N=2) | DB Period: Setmelanotide 25 mg QW (N=1) | DB Period: Setmelanotide 3 mg QD (N=9) | DB Period: Setmelanotide 30 mg QW (N=7) | OL Period: Setmelanotide 20 mg QW (N=1) | OL Period: Setmelanotide 25 mg QW (N=1) | OL Period: Setmelanotide 30 mg QW (N=14)
Injection site erythema (General disorders) | 0 | 0 | 1 | 1 | 1 | 4 | 2 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 0 | 1 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Injection site mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05194124/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT05194124/SAP_001.pdf